CLINICAL TRIAL: NCT06371209
Title: Validating Normal Kinematic Motion in Residual Limb Musculature of Ewing Amputees
Brief Title: Kinematics of Ewing Amputees
Status: Enrolling by invitation | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Matthew Carty, Director, Lower Extremity Transplant Program, Brigham and Women's Hospital, Brigham and Women's Hospital
Other Study IDs: 2022P000619
Record Dates: First submitted 2023-12-05; First posted 2024-04-17 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Lower Extremity Amputation; Trans-Tibial Amputation; Traumatic Lower Extremity Amputation; Agonist-Antagonist Myoneural Interface
Keywords: Amputation; Kinematics; Gait

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Ewing Amputees: Amputees who have previously undergone Agonist-Antagonist Myoneural Interface construction at the trans-tibial level
  Interventions: Procedure: Modified Amputation
- Standard Amputees: Amputees who have previously undergone trans-tibial level amputations without the construction of Agonist-Antagonist Myoneural Interfaces
  Interventions: Procedure: Standard Amputation

INTERVENTIONS:
Procedure: Modified Amputation — Modified amputation procedure
  Groups: Ewing Amputees
Procedure: Standard Amputation — Standard amputation procedure
  Groups: Standard Amputees

SUMMARY:
The agonist-antagonist myoneural interface (AMI) construct, known as the Ewing amputation at the trans-tibial level, has been shown to create a bi-directional neural communication platform as a means of controlling and interpreting proprioceptive feedback from a prosthetic joint. In AMI constructs, agonist-antagonist muscles are mechanically coupled within the residual limb, and volitional contraction of an agonist passively stretches that muscle's antagonist. The natural neural responses from muscle spindles within both muscles are then interpreted by the central nervous system as sensations of joint position and speed, associated with movement of the prosthesis.

The aim of this research protocol is to evaluate the electromyographic and kinematic patterns of participants who have undergone unilateral lower extremity Ewing Amputation in order to determine how similar their residual limb data is when compared to their intact limb data. A secondary aim of this research may include comparison of the Ewing participant cohort's biomechanical patterns to a similar cohort of participants who have undergone standard amputation.

The investigators hypothesize that the affected limb of patients with the Ewing procedure will demonstrate a pattern of electromyographic activation of their AMI constructs and kinematic data that recapitulates the pattern seen in their intact limb. The investigators secondarily hypothesize that the kinematic assessment of Ewing Amputation patients will demonstrate patterns that are significantly more physiologic than those witnessed in similar assessments of standard amputees.

DETAILED DESCRIPTION:
The specific aim of this research protocol is to evaluate the electromyographic and kinematic patterns of participants who have undergone unilateral lower extremity Ewing Amputation in order to determine how similar their residual limb data is when compared to their intact limb data. A secondary aim of this research may include comparison of the Ewing participant cohort's biomechanical patterns to a similar cohort of participants who have undergone standard amputation.

The investigators hypothesize that the affected limb of participants with the Ewing procedure will demonstrate a pattern of electromyographic activation of their AMI constructs and kinematic data that recapitulates the pattern seen in their intact limb. The investigators secondarily hypothesize that the kinematic assessment of Ewing Amputation participants will demonstrate patterns that are significantly more physiologic than those witnessed in similar assessments of standard amputees.

This will be a cross-sectional study with only one visit. A convenience sample of 16 participants who have previously undergone a lower extremity Ewing amputation will be recruited for the proposed study. Participants may subsequently be matched with up to 16 control participants who have previously undergone standard amputation procedures.

Participants will be assessed in a single session in the Motion Analysis Lab (MAL) at Spaulding Rehabilitation Hospital (SRH). Each visit will consist of the procedures described below and is expected to last about two and a half (2.5) hours.

The investigators will collect demographic data for each participant to help with the study population characterization. Such data will include questions about past medical and surgical history, height, weight, and prosthetic and functional history. In addition to self-reported data from the participant, the investigators may review the electronic medical record of any Mass General Brigham (MGB) participant in order to confirm demographic information.

Clinical tests may be conducted by the investigators to assess participant's lower extremities. Clinical tests may include functional examination of each participant's range of motion (ROM) and muscular strength for the lower extremities. Passive hip movements (flexion, abduction, adduction, internal and external rotation), knee flexion and extension, and ankle dorsiflexion and plantar flexion may be assessed with a goniometer if the joint is present for each limb.

Gait evaluations will be performed in the MAL during one session. Participants will be asked to change into shorts and a short-sleeved shirt (such articles of clothing can be provided by the lab if needed). Data will be gathered simultaneously with an electromyographic (EMG) system and a motion capture system. Both systems are part of SRH inventory and are routinely used in clinical care.

The spatio-temporal parameters, kinematic data and electromyographic data obtained from the Motion Capture System are the primary outcomes. As an exploratory analysis, the investigators will seek the possibility of assessing other items such as symmetry measurements and energy recovery as secondary outcomes.

Biomechanical data will be collected to study gait patterns. To ensure the accuracy of the biomechanical data, the investigators may gather additional data on the participant's gait patterns using a ten-camera motion analysis system (VICON) that is equipped with force plates (AMTI). To track participant movement, reflective markers will be attached using bio-adhesive tape to the participant's lower limbs and trunk based on anatomical landmarks (for example: second metatarsal head, center of calcaneus, lateral malleolus, lateral shank, distal lateral epicondyles, lateral thigh, anterior superior iliac spine, and the sacrum). Reflective markers may also be placed on the prosthesis to track its movement. The VICON system includes standard video cameras to record the session. The investigators will ask study participants permission to video record the gait trials and use the material for scientific presentations.

Electromyographic (EMG) data may be collected to study the characteristics of lower extremity muscle activation patterns during gait. The investigators will follow the Surface Electromyography for the Non-Invasive Assessment of Muscles (SENIAM) guidelines to place electrodes on several lower extremity muscles. Those may include the following: gastrocnemius, tibialis anterior, peroneal longus, rectus femoris, vastus lateralis, biceps femoris, or gluteus maximus. EMG electrodes will be attached using bio-adhesive double-sided tape and secured with Coban (self-adherent wrap) if needed. Portable ultrasonography may be used to localize muscles for proper electrode placement at this time. To ensure proper contact, the skin will be prepped for the electrodes; the area will be cleaned with alcohol swabs and shaved if necessary. Data from the electrodes will be gathered simultaneously with an acquisition system synchronized with the motion analysis system.

In the event that the surface EMG (sEMG) is not sufficiently robust to carry out the trials, the investigators will move to needle-based electrodes. If it is determined that needle-based electrodes are to be used to collect EMG data on the residual limb of a given participant, the amputee participant will meet with a clinician on the protocol with significant experience working with placement of electrodes in residual limb musculature. Since the musculature on the residual limb will be different for each participant, the participants will be instructed to make test contractions (e.g. ankle dorsiflexion or plantarflexion) to assist in localizing muscle sites. Sterile fine-wire electrodes will then be placed by the clinician on the protocol in each of the muscles of interest. The needles for electrode placement are 27-gauge needles. These needles are used acutely in the clinical space to insert the fine-wire electrodes into the muscles. The needles are then removed, leaving behind the fine-wire electrode. The fine-wire electrode is extremely fine, with a diameter of .051 mm. Because electrode placement is minimally invasive, this will occur at the gait lab.

Each participant will be asked to complete gross motor task assessing static and dynamic balance in their shoes and with the prosthetic device they typically wear for community ambulation. The participant will be asked to do this several times until 5-10 trials with good foot contacts onto the force plates are collected for each side (leg) of the body. There will be regular rest breaks during testing. At the end of the session, a trained study investigator will perform a brief visual check of the areas where the surface electrodes were in contact with the skin to assess these pressure areas. This will mark the end of the study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral lower extremity amputees
* Greater than 12 months post-amputation procedure
* Possession and use of a working prosthesis as determined by subject's ability to wear it for 8 hours daily
* A stable, well-fitting socket as indicated by no prosthetic modifications within the prior 14 days and no plans to modify it within the following 30 days
* Follow-up visit with their prosthetist within the past 3 months
* The ability to walk independently without an assistive device
* The ability to follow directions and communicate pain or discomfort

Exclusion Criteria:

* Patients beyond the stated age restrictions will be excluded
* Patients who have any underlying neurologic, orthopedic, or cardiopulmonary impairment that affects their gait as assessed by the study clinician.
* Patients with any medical or functional limitations preventing them from ambulating safely and independently without an assistive device.
* Patients will be excluded who do not have a prosthesis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Trans-tibial amputees local to or visiting the Massachusetts area
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2022-05-17 (Actual); Primary Completion 2026-06-29 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Duration of co-contraction of the ankle dorsi/plantar-flexor muscles during gait | Baseline
  The percentage of the gait cycle during which both the Tibialis Anterior and the Gastrocnemius muscles are active is estimated for the residuum and the contralateral side.
Symmetry of duration of co-contraction of the ankle dorsi/plantar-flexor muscles during gait | Baseline
  This is estimated by calculating the difference between the duration of co-contraction for the residuum and for the contralateral limb.

SECONDARY OUTCOMES:
Symmetry of ankle power generation | Baseline
  This is estimated by calculating the difference between the peak ankle power generation on the affected side (i.e., prosthesis side) and the contralateral limb.
Symmetry of peak knee flexion during stance | Baseline
  This is estimated by calculating the difference between the peak knee flexion for the residuum and for the contralateral limb.

OTHER OUTCOMES:
Symmetry of step length | Baseline
  This is estimated by calculating the difference in step length between the affected side (i.e., prosthesis side) step length and the contralateral limb step length.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Carty, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Mass General Brigham, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No plan for individual participant data sharing

REFERENCES:
- [Background] Srinivasan SS, Diaz M, Carty M, Herr HM. Towards functional restoration for persons with limb amputation: A dual-stage implementation of regenerative agonist-antagonist myoneural interfaces. Sci Rep. 2019 Feb 13;9(1):1981. doi: 10.1038/s41598-018-38096-z. PMID 30760764
- [Background] Clites TR, Carty MJ, Ullauri JB, Carney ME, Mooney LM, Duval JF, Srinivasan SS, Herr HM. Proprioception from a neurally controlled lower-extremity prosthesis. Sci Transl Med. 2018 May 30;10(443):eaap8373. doi: 10.1126/scitranslmed.aap8373. PMID 29848665
- [Background] Srinivasan SS, Carty MJ, Calvaresi PW, Clites TR, Maimon BE, Taylor CR, Zorzos AN, Herr H. On prosthetic control: A regenerative agonist-antagonist myoneural interface. Sci Robot. 2017 May 31;2(6):eaan2971. doi: 10.1126/scirobotics.aan2971. PMID 33157872
- [Background] Clites TR, Carty MJ, Srinivasan S, Zorzos AN, Herr HM. A murine model of a novel surgical architecture for proprioceptive muscle feedback and its potential application to control of advanced limb prostheses. J Neural Eng. 2017 Jun;14(3):036002. doi: 10.1088/1741-2552/aa614b. Epub 2017 Feb 17. PMID 28211795
- [Background] Clites TR, Herr HM, Srinivasan SS, Zorzos AN, Carty MJ. The Ewing Amputation: The First Human Implementation of the Agonist-Antagonist Myoneural Interface. Plast Reconstr Surg Glob Open. 2018 Nov 16;6(11):e1997. doi: 10.1097/GOX.0000000000001997. eCollection 2018 Nov. PMID 30881798
- [Background] Ziegler-Graham K, MacKenzie EJ, Ephraim PL, Travison TG, Brookmeyer R. Estimating the prevalence of limb loss in the United States: 2005 to 2050. Arch Phys Med Rehabil. 2008 Mar;89(3):422-9. doi: 10.1016/j.apmr.2007.11.005. PMID 18295618
- [Background] Brown BJ, Iorio ML, Klement M, Conti Mica MR, El-Amraoui A, O'Halloran P, Attinger CE. Outcomes after 294 transtibial amputations with the posterior myocutaneous flap. Int J Low Extrem Wounds. 2014 Mar;13(1):33-40. doi: 10.1177/1534734614520706. Epub 2014 Feb 6. PMID 24510319